CLINICAL TRIAL: NCT03467932
Title: A Placebo-controlled, Multi-center, Randomized, Phase 2b Study to Evaluate the Efficacy and Safety of ORMD-0801 in Type 2 Diabetes Mellitus Patients With Inadequate Glycemic Control on Oral Therapy
Brief Title: A Study to Evaluate the Efficacy and Safety of ORMD-0801 (Oral Insulin) in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oramed, Ltd. (Industry)
Collaborators: Integrium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORA-D-015
Record Dates: First submitted 2018-03-01; First posted 2018-03-16 (Actual); Results first posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: T2DM (Type 2 Diabetes Mellitus)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin; Edetic Acid; Fish Oils; Silicon Dioxide; Polysorbates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Single-Blind Placebo Run-in (Masking will be with Participant):
  During the placebo run-in period, subjects will self-administer blinded placebo study medication at night prior to bedtime (@10 PM ± 90 min. each night, no sooner than 2 hrs. after dinner). Outpatient glycemic levels and adverse events will be measured using self-monitored blood glucose (SMBG) and recorded in a diary. Treatment Period (Masking: Participant, Care Provider, Investigator, Outcomes Assessor) There are 2 Cohorts, A and B.
  Part 1 In the first 2 weeks of active treatment, subjects will receive double-blind therapy according to their randomized regimen (placebo or ORMD-0801) to be taken QHS (bedtime), BID (2 X / day) or TID.
  Part 2 Subjects will remain on fixed doses of ORMD-0801 or matched placebo for 10 weeks. Doses will not be adjusted unless clinically indicated for adverse events or hypoglycemia. Treatment arms will consist of subjects receiving ORMD-0801 QHS, BID, and TID versus placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Cohort A: ORMD-0801 once daily - QHS (Active Comparator): Dosed in the evening prior to bedtime (@ 10 PM ± 90 minutes)
  Interventions: Drug: Cohort A: ORMD-0801
- Cohort A: ORMD-0801 twice daily - BID (Active Comparator): Dosed in the evening prior to bedtime (@ 10 PM ± 90 minutes) and 30-45 minutes prior to breakfast.
  Interventions: Drug: Cohort A: ORMD-0801
- Cohort A: ORMD-0801 three times daily - TID (Active Comparator): ORMD-0801 three times daily - TID: dosed in the evening prior to bedtime (@ 10 PM ± 90 minutes) and 30-45 minutes prior to breakfast and lunch.
  Interventions: Drug: Cohort A: ORMD-0801
- Cohort A: Matched Placebo Oral Capsule (Placebo Comparator): Placebo matched to one of the three active comparator arms. (either QHS, BID, or TID)
  Interventions: Drug: Placebo oral capsule
- Cohort A: Excipient-Matched Placebo three times daily-TID (Placebo Comparator): Excipient matched placebo in a non-randomized single-blind fashion, TID, dosed in the evening prior to bedtime (@ 10 PM ± 90 minutes) and 30-45 minutes prior to breakfast and lunch.
  This is an exploratory arm, per FDA. The results of this arm are not included in the primary analysis.
  Interventions: Drug: Placebo oral capsule
- Cohort B:ORMD-0801, 8 mg once daily - QHS: (Active Comparator): ORMD-0801 8 mg once daily - QHS: dosed in the evening prior to bedtime (@ 10 PM ± 90 minutes)
  Interventions: Drug: Cohort B: ORMD-0801
- Cohort B: ORMD-0801 8 mg twice daily - BID (Active Comparator): ORMD-0801 8 mg twice daily - BID: dosed in the evening prior to bedtime (@ 10 PM ± 90 minutes) and 30-45 minutes prior to breakfast.
  Interventions: Drug: Cohort B: ORMD-0801
- Cohort B: ORMD-0801 16 mg once daily - QHS: (Active Comparator): ORMD-0801 16 mg once daily - QHS: dosed in the evening prior to bedtime (@ 10 PM ± 90 minutes)
  Interventions: Drug: Cohort B: ORMD-0801
- Cohort B: ORMD-0801 16 mg twice daily - BID (Active Comparator): ORMD-0801 16 mg twice daily - BID: dosed in the evening prior to bedtime (@ 10 PM ± 90 minutes) and 30-45 minutes prior to breakfast.
  Interventions: Drug: Cohort B: ORMD-0801
- Cohort B - Matched Placebo Oral Capsule (Placebo Comparator): Cohort B - Matched Placebo Oral Capsule: dosed in the evening prior to bedtime (@ 10 PM ± 90 minutes)
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Cohort A: ORMD-0801 — Part 1 In the first two weeks of active treatment (Part 1) subjects will receive double-blind therapy according to their randomized regimen (placebo or ORMD-0801) to be taken QHS, BID or TID. Subjects will undergo a step-wise dose escalation from a starting dose of 16 mg (Visit 3), to 24 mg (Visit 4), to a top dose of 32 mg (Visit 5 onward). Subjects will then enter Part 2.
  Part 2:
  During Part 2, subjects will remain on fixed doses of ORMD-0801 (or matched placebo) for 10 weeks. Doses will not be adjusted unless clinically indicated for adverse events or hypoglycemia.
  Other Names: Oral Insulin
  Arms: Cohort A: ORMD-0801 once daily - QHS; Cohort A: ORMD-0801 three times daily - TID; Cohort A: ORMD-0801 twice daily - BID
Drug: Placebo oral capsule — Placebo provided QHS, BID, TID
  Other Names: SBTI, disodium EDTA, fish oil, aerosil, and TWEEN 80.
  Arms: Cohort A: Excipient-Matched Placebo three times daily-TID; Cohort A: Matched Placebo Oral Capsule; Cohort B - Matched Placebo Oral Capsule
Drug: Cohort B: ORMD-0801 — Part 1 In the first two weeks of active treatment, subjects will receive double-blind therapy according to their randomized regimen (ORMD 0801 8 mg or 16 mg, or matched placebo) to be taken QHS or BID. Subjects will then enter Part 2 at the same dose and regimen administered in Part 1.
  Part 2 Subjects will remain on fixed doses of ORMD-0801 (or matched placebo) for 10 weeks. Doses will not be adjusted unless clinically indicated for adverse events or hypoglycemia.
  Other Names: Oral Insulin
  Arms: Cohort B: ORMD-0801 16 mg once daily - QHS:; Cohort B: ORMD-0801 16 mg twice daily - BID; Cohort B: ORMD-0801 8 mg twice daily - BID; Cohort B:ORMD-0801, 8 mg once daily - QHS:

SUMMARY:
This is a four-way (Participant, Care Provider, Investigator, Outcomes Assessor) masked (blinded) study designed to explore the efficacy of ORMD-0801 when given in different regimens across a dose range for up to 12 weeks in subjects with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
This study is designed to explore the efficacy of ORMD-0801 when given in different regimens across a dose range for up to 12 weeks in subjects with type 2 diabetes mellitus (T2DM). There are two cohorts in this study. Approximately 360 subjects with T2DM will initially undergo a 2-week, single-blind placebo run-in period (Visits 1 and 2), followed by a 12-week treatment period (Visits 3 through 9). Cohort A will enroll 285 subjects; Cohort B will enroll 75 subjects

For 265 of the 285 subjects of Cohort A, the total 12-week treatment period will include a Part 1"dose escalation" interval (2 weeks, Visits 3 and 4) and a Part 2 stable dose "maintenance" interval (10 weeks, Visits 5 through 9).

In addition, per FDA request, the remaining 20 subjects (of the cohort total of 285 enrolled subjects) will receive excipient-matched placebo in a non-randomized single-blind fashion, TID (3 times per day), according to the same schedule as described above.

For Cohort B (75 of the 360 total subjects), the total 12-week treatment period will include a stable dosing period for both Part 1 (2 weeks, Visits 3 and 4) and Part 2 (10 weeks, Visits 5 through 9).

Cohort A data will be analyzed after Cohort A data collection has been completed (last subject for Cohort A screened on 7 May 2019). Estimated completion for Cohort A is October 2019. Cohort B data will be analyzed following the release of results from Cohort A.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 and older.
* Established diagnosis of T2DM for at least 6 months prior to Screening, with an HbA1C (glycated hemoglobin) ≥ 7.5%.
* Stable dose of metformin (at least 1500 mg or maximally tolerated dose)/oral antidiabetic (OAD) for a period of at least 3 months prior to screening.
* Taking metformin only or metformin in addition to no more than two of the following: DPP-4 (DiPeptidyl Peptidase-4), SGLT-2 (Sodium-GLucose coTransporter-2), or TZD (Thiazolidinediones).
* Body mass index (BMI) of up to 40 kg/m2 at Screening and stable weight, with no more than 5 kg gain or loss in the 3 months prior to Screening.
* Renal function - eGFR (estimated glomerular filtration rate) > 30 ml/min/1.73 m2
* Females of childbearing potential must have a negative serum pregnancy test result at Screening.

Exclusion Criteria:

* Subjects with insulin-dependent diabetes

  1. has a history of type 1 diabetes mellitus or a history of ketoacidosis, or subject is assessed by the investigator as possibly having type 1 diabetes mellitus confirmed by a C-peptide <0.7 ng/mL (0.23 nmol/L).
  2. has a history of other specific types of diabetes (e.g., genetic syndromes, secondary pancreatic diabetes, diabetes due to endocrinopathies, drug- or chemical-induced, and post-organ transplant).
* Treatment with glucosidase inhibitor, insulin secretagogues (other than sulfonylureas), glucagon-like peptide 1 (GLP-1) agonists within 3 months prior to Visit 1.
* History of any basal, pre-mix or prandial insulin (greater than 7 days) within 6 months prior to Screening.
* History of >2 episodes of severe hypoglycemia within 6 months prior to Screening.
* History of hypoglycemic unawareness (episodes of severe hypoglycemia with seizure or requiring third-party intervention or documented low blood glucose without associated autonomic symptoms)
* Subjects with the following secondary complications of diabetes:

  1. Active proliferative retinopathy as confirmed by a dilated ophthalmoscopy/retinal photography examination performed (by a qualified person as per the country legislation) within 6 months prior to Screening.
  2. Renal dysfunction: eGFR < 30 ml/min/1.73 m2
  3. History of proliferative retinopathy or severe form of neuropathy or cardiac autonomic neuropathy (CAN)
  4. Uncontrolled or untreated severe hypertension defined as systolic blood pressure above or equal to 180 mmHg and/or diastolic blood pressure above or equal to 120 mmHg
  5. Presence of unstable angina or myocardial infarction within 6 months prior to Screening, Grade 3 or 4 congestive heart failure (CHF) according to the New York Heart Association (NYHA) criteria, valvular heart disease, cardiac arrhythmia requiring treatment, pulmonary hypertension, cardiac surgery, history/occurrence of coronary angioplasty and/or stroke or transient ischemic attack (TIA) within 6 months prior to Screening.
* Subjects with psychiatric disorders which, per investigator judgment may have an impact on the safety of the subject or interfere with the subject's participation or compliance in the study.
* Subjects who needed (in the last 12 months) or may require systemic (oral, intravenous, intramuscular) glucocorticoid therapy for more than 2 weeks during the study period.
* 9. Laboratory abnormalities at Screening include:

  1. C-peptide < 1.0 ng/mL
  2. Abnormal serum thyrotropin (TSH) levels below the lower limit of normal or >1.5X the upper limit of normal
  3. Elevated liver enzymes (alanine transaminase (ALT), alanine aminotransferase (AST), alkaline phosphatase) >2X the upper limit of normal.
  4. Very high triglyceride levels (>600 mg/dL); a single repeat test is allowable.
  5. Any relevant abnormality that would interfere with the efficacy or the safety assessments during the study treatment administration.
* Positive history of active liver disease (other than non-alcoholic hepatic steatosis), including chronic hepatitis B or C, primary biliary cirrhosis, or active symptomatic gallbladder disease.
* Positive history of HIV.
* Use of the following medications:

  1. History of any basal, pre-mix or prandial insulin (greater than 7 days) within 6 months prior to Screening.
  2. Administration of thyroid preparations or thyroxine (except in subjects on stable replacement therapy) within 6 weeks prior to Screening.
  3. Administration of systemic long-acting corticosteroids within two months or prolonged use (more than one week) of other systemic corticosteroids or inhaled corticosteroids (if daily dosage is > 1,000 μg equivalent beclomethasone) within 30 days prior to Screening. Intra-articular and/or topical corticosteroids are not considered systemic.
  4. Use of medications known to modify glucose metabolism or to decrease the ability to recover from hypoglycemia such as oral, parenteral, and inhaled steroids (as discussed above), and immunosuppressive or immunomodulating agents.
* Known allergy to soy.
* Subject is on a weight loss program and is not in the maintenance phase or subject has started weight loss medication (e.g., orlistat or liraglutide), within 8 weeks prior to Screening.
* Subject has had bariatric surgery.
* Subject is pregnant or breastfeeding.
* Subject is a user of recreational or illicit drugs or has had a recent history (within 1 year of Screening) of drug or alcohol abuse or dependence. (Note: Alcohol abuse includes heavy alcohol intake as defined by >3 drinks per day or >14 drinks per week, or binge drinking) at Screening. Occasional intermittent use of cannabinoid products will be allowed provided that no cannabinoid products have been used during the 1 week prior to each visit.
* One or more contraindications to metformin as per local label.
* History of gastrointestinal disorders (e.g. hypochlorhydria) with the potential to interfere with drug absorption.
* At the Principal Investigator's discretion, any condition or other factors that are deemed unsuitable for subject enrollment into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2020-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel M Neutel, M. D., Principal Investigator — Orange County Research Center
Locations (1):
- AA MRC, Flint, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited into two primary Cohorts, A and B.
  Cohort A:
  1. ORMD-0801 1X daily
  2. ORMD-0801 2X daily
  3. ORMD-0801 3X daily
  4. Matched Placebo
  Sub-Cohort A 20 subjects Per FDA, excipient matched placebo; randomized single-blind, TID, same schedule as for Cohort A.
  Not part of primary analysis.
  Cohort B:
  1. ORMD-0801 8 mg 1X daily
  2. ORMD-0801 8 mg 2X daily
  3. ORMD-0801 16 mg 1X daily
  4. ORMD-0801 16 mg 2X daily
  5. Excipient matched placebo once daily
Pre-assignment Details: After screening, patients underwent a 2-week, single-blind placebo run-in period (Visits 1[baseline] and 2), followed by a 12-week treatment period.
  Cohort A:
  12-wk treatment period, 2 parts. Part 1, dose escalation interval for 2 weeks (Visits 3 and 4) Part 2, stable dose "maintenance" for 10 weeks (Visits 5-9).
  ;
  Cohort B:
  12-wk treatment period, 2 parts. Part 1, stable dosing for 2 weeks (Visits 3 and 4) Part 2, stable dosing for 10 weeks, Visits 5-9).
Groups:
- Cohort A: ORMD-0801 Once Daily - QHS: Dosed in the evening prior to bedtime (@ 10 PM ± 90 minutes)
  Cohort A: ORMD-0801: Part 1 In the first two weeks of active treatment (Part 1) subjects will receive double-blind therapy according to their randomized regimen (placebo or ORMD-0801) to be taken QHS, BID or TID. Subjects will undergo a step-wise dose escalation from a starting dose of 16 mg (Visit 3), to 24 mg (Visit 4), to a top dose of 32 mg (Visit 5 onward). Subjects will then enter Part 2.
  Part 2:
  During Part 2, subjects will remain on fixed doses of ORMD-0801 (or matched placebo) for 10 weeks. Doses will not be adjusted unless clinically indicated for adverse events or hypoglycemia.
- Cohort A: ORMD-0801 Twice Daily - BID: Dosed in the evening prior to bedtime (@ 10 PM ± 90 minutes) and 30-45 minutes prior to breakfast.
  Cohort A: ORMD-0801: Part 1 In the first two weeks of active treatment (Part 1) subjects will receive double-blind therapy according to their randomized regimen (placebo or ORMD-0801) to be taken QHS, BID or TID. Subjects will undergo a step-wise dose escalation from a starting dose of 16 mg (Visit 3), to 24 mg (Visit 4), to a top dose of 32 mg (Visit 5 onward). Subjects will then enter Part 2.
  Part 2:
  During Part 2, subjects will remain on fixed doses of ORMD-0801 (or matched placebo) for 10 weeks. Doses will not be adjusted unless clinically indicated for adverse events or hypoglycemia.
- Cohort A: ORMD-0801 Three Times Daily - TID: ORMD-0801 three times daily - TID: dosed in the evening prior to bedtime (@ 10 PM ± 90 minutes) and 30-45 minutes prior to breakfast and lunch.
  Cohort A: ORMD-0801: Part 1 In the first two weeks of active treatment (Part 1) subjects will receive double-blind therapy according to their randomized regimen (placebo or ORMD-0801) to be taken QHS, BID or TID. Subjects will undergo a step-wise dose escalation from a starting dose of 16 mg (Visit 3), to 24 mg (Visit 4), to a top dose of 32 mg (Visit 5 onward). Subjects will then enter Part 2.
  Part 2:
  During Part 2, subjects will remain on fixed doses of ORMD-0801 (or matched placebo) for 10 weeks. Doses will not be adjusted unless clinically indicated for adverse events or hypoglycemia.
- Cohort A (Sub-Cohort A): Excipient-Matched Placebo Three Times Daily-TID: Excipient matched placebo in a non-randomized single-blind fashion, TID, dosed in the evening prior to bedtime (@ 10 PM ± 90 minutes) and 30-45 minutes prior to breakfast and lunch.
  Placebo oral capsule: Placebo provided QHS, BID, TID
  Per FDA, this sub-Cohort A is an exploratory endpoint, and not part of the primary analysis.
- Cohort B:ORMD-0801, 8 mg Once Daily - QHS:: ORMD-0801 8 mg once daily - QHS: dosed in the evening prior to bedtime (@ 10 PM ± 90 minutes)
  Cohort B: ORMD-0801: Part 1 In the first two weeks of active treatment, subjects will receive double-blind therapy according to their randomized regimen (ORMD 0801 8 mg or 16 mg, or matched placebo) to be taken QHS or BID. Subjects will then enter Part 2 at the same dose and regimen administered in Part 1.
  Part 2 Subjects will remain on fixed doses of ORMD-0801 (or matched placebo) for 10 weeks. Doses will not be adjusted unless clinically indicated for adverse events or hypoglycemia.
- Cohort B: ORMD-0801 8 mg Twice Daily - BID: ORMD-0801 8 mg twice daily - BID: dosed in the evening prior to bedtime (@ 10 PM ± 90 minutes) and 30-45 minutes prior to breakfast.
  Cohort B: ORMD-0801: Part 1 In the first two weeks of active treatment, subjects will receive double-blind therapy according to their randomized regimen (ORMD 0801 8 mg or 16 mg, or matched placebo) to be taken QHS or BID. Subjects will then enter Part 2 at the same dose and regimen administered in Part 1.
  Part 2 Subjects will remain on fixed doses of ORMD-0801 (or matched placebo) for 10 weeks. Doses will not be adjusted unless clinically indicated for adverse events or hypoglycemia.
- Cohort B: ORMD-0801 16 mg Once Daily - QHS:: ORMD-0801 16 mg once daily - QHS: dosed in the evening prior to bedtime (@ 10 PM ± 90 minutes)
  Cohort B: ORMD-0801: Part 1 In the first two weeks of active treatment, subjects will receive double-blind therapy according to their randomized regimen (ORMD 0801 8 mg or 16 mg, or matched placebo) to be taken QHS or BID. Subjects will then enter Part 2 at the same dose and regimen administered in Part 1.
  Part 2 Subjects will remain on fixed doses of ORMD-0801 (or matched placebo) for 10 weeks. Doses will not be adjusted unless clinically indicated for adverse events or hypoglycemia.
- Cohort B: ORMD-0801 16 mg Twice Daily - BID: ORMD-0801 16 mg twice daily - BID: dosed in the evening prior to bedtime (@ 10 PM ± 90 minutes) and 30-45 minutes prior to breakfast.
  Cohort B: ORMD-0801: Part 1 In the first two weeks of active treatment, subjects will receive double-blind therapy according to their randomized regimen (ORMD 0801 8 mg or 16 mg, or matched placebo) to be taken QHS or BID. Subjects will then enter Part 2 at the same dose and regimen administered in Part 1.
  Part 2 Subjects will remain on fixed doses of ORMD-0801 (or matched placebo) for 10 weeks. Doses will not be adjusted unless clinically indicated for adverse events or hypoglycemia.
Period: Overall Study
Arm/Group | Cohort A: ORMD-0801 Once Daily - QHS | Cohort A: ORMD-0801 Twice Daily - BID | Cohort A: ORMD-0801 Three Times Daily - TID | Cohort A: Matched Placebo Oral Capsule | Cohort A (Sub-Cohort A): Excipient-Matched Placebo Three Times Daily-TID | Cohort B:ORMD-0801, 8 mg Once Daily - QHS: | Cohort B: ORMD-0801 8 mg Twice Daily - BID | Cohort B: ORMD-0801 16 mg Once Daily - QHS: | Cohort B: ORMD-0801 16 mg Twice Daily - BID | Cohort B - Matched Placebo Oral Capsule
Started | 69 | 68 | 69 | 66 | 20 | 15 | 17 | 18 | 15 | 16
Completed | 62 | 58 | 58 | 56 | 19 | 13 | 15 | 16 | 11 | 14
Not Completed | 7 | 10 | 11 | 10 | 1 | 2 | 2 | 2 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Cohort A+Cohort B Combined: Matched Oral Capsule Placebo: Placebo matched to one of the three active comparator arms. (either QHS, BID, or TID)
  Placebo oral capsule: Placebo provided QHS, BID, TID
  This combined arm does not include the sub-cohort A, Excipient-Matched Placebo which per FDA is an exploratory endpoint, not part of the primary analysis.
- Cohort A: ORMD-0801 Once Daily - QD: Dosed in the evening prior to bedtime (@ 10 PM ± 90 minutes)
  Cohort A: ORMD-0801: Part 1 In the first two weeks of active treatment (Part 1) subjects will receive double-blind therapy according to their randomized regimen (placebo or ORMD-0801) to be taken QHS, BID or TID. Subjects will undergo a step-wise dose escalation from a starting dose of 16 mg (Visit 3), to 24 mg (Visit 4), to a top dose of 32 mg (Visit 5 onward). Subjects will then enter Part 2.
  Part 2:
  During Part 2, subjects will remain on fixed doses of ORMD-0801 (or matched placebo) for 10 weeks. Doses will not be adjusted unless clinically indicated for adverse events or hypoglycemia.
- Cohort B:ORMD-0801, 8 mg Once Daily - QD: ORMD-0801 8 mg once daily - QHS: dosed in the evening prior to bedtime (@ 10 PM ± 90 minutes)
  Cohort B: ORMD-0801: Part 1 In the first two weeks of active treatment, subjects will receive double-blind therapy according to their randomized regimen (ORMD 0801 8 mg or 16 mg, or matched placebo) to be taken QHS or BID. Subjects will then enter Part 2 at the same dose and regimen administered in Part 1.
  Part 2 Subjects will remain on fixed doses of ORMD-0801 (or matched placebo) for 10 weeks. Doses will not be adjusted unless clinically indicated for adverse events or hypoglycemia.
- Cohort B: ORMD-0801 16 mg Once Daily - QD: ORMD-0801 16 mg once daily - QHS: dosed in the evening prior to bedtime (@ 10 PM ± 90 minutes)
  Cohort B: ORMD-0801: Part 1 In the first two weeks of active treatment, subjects will receive double-blind therapy according to their randomized regimen (ORMD 0801 8 mg or 16 mg, or matched placebo) to be taken QHS or BID. Subjects will then enter Part 2 at the same dose and regimen administered in Part 1.
  Part 2 Subjects will remain on fixed doses of ORMD-0801 (or matched placebo) for 10 weeks. Doses will not be adjusted unless clinically indicated for adverse events or hypoglycemia.
- Sub-Cohort A: Excipient Matched Placebo: Data collected from participants who received excipient-matched placebo was an exploratory efficacy evaluation and therefore excluded from the primary and secondary analysis.
- Total: Total of all reporting groups
Arm/Group | Cohort A+Cohort B Combined: Matched Oral Capsule Placebo | Cohort A: ORMD-0801 Once Daily - QD | Cohort A: ORMD-0801 Twice Daily - BID | Cohort A: ORMD-0801 Three Times Daily - TID | Cohort B:ORMD-0801, 8 mg Once Daily - QD | Cohort B: ORMD-0801 8 mg Twice Daily - BID | Cohort B: ORMD-0801 16 mg Once Daily - QD | Cohort B: ORMD-0801 16 mg Twice Daily - BID | Sub-Cohort A: Excipient Matched Placebo | Total
Number analyzed (Participants) | 82 | 69 | 68 | 69 | 15 | 17 | 18 | 15 | 20 | 373
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.92 (9.914) | 56.72 (10.766) | 55.68 (10.569) | 55.22 (11.663) | 53.66 (8.22) | 56.87 (9.132) | 54.98 (11.229) | 54.98 (11.785) | 64.08 (9.218) | 55.73 (10.544)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 27 | 23 | 29 | 5 | 7 | 7 | 4 | 8 | 143
  Male | 49 | 42 | 45 | 40 | 10 | 10 | 11 | 11 | 12 | 230
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48 | 36 | 37 | 36 | 9 | 8 | 9 | 8 | 0 | 191
  Not Hispanic or Latino | 33 | 32 | 29 | 33 | 6 | 6 | 9 | 6 | 20 | 174
  Unknown or Not Reported | 1 | 1 | 2 | 0 | 0 | 3 | 0 | 1 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 2 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 4
  Black or African American | 11 | 7 | 8 | 8 | 3 | 4 | 1 | 1 | 3 | 46
  White | 69 | 59 | 57 | 58 | 12 | 11 | 16 | 11 | 17 | 310
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 6
BMI [Mean (Standard Deviation); unit: Kg/M^2] | 31.137 (4.7750) | 31.721 (4.9409) | 30.447 (4.7710) | 31.191 (4.0045) | 31.759 (4.4393) | 31.005 (5.0333) | 31.881 (6.0514) | 30.776 (5.4530) | 31.310 (5.5976) | 31.171 (4.7203)
HbA1c [Mean (Standard Deviation); unit: percent HbA1c] | 9.46 (1.434) | 8.96 (1.281) | 9.36 (1.656) | 9.64 (1.578) | 9.83 (1.759) | 8.46 (1.104) | 8.96 (1.420) | 9.18 (1.687) | 8.93 (0.929) | 9.31 (1.512)
Diabetes Medications [Count of Participants; unit: Participants]
  Metformin Alone | 22 | 20 | 20 | 12 | 6 | 5 | 7 | 5 | 6 | 103
  Metformin, No Sulfonylureas, but At Least 1 Other Medication | 13 | 10 | 8 | 12 | 1 | 0 | 1 | 2 | 1 | 48
  Metformin with Sulfonylureas Only | 33 | 30 | 26 | 33 | 7 | 7 | 8 | 3 | 4 | 151
  Metformin with Sulfonylureas and Other Medication(s) | 10 | 5 | 8 | 6 | 0 | 1 | 1 | 3 | 6 | 40
  Not on Metformin, But On 1 Other Medication | 4 | 4 | 3 | 4 | 1 | 2 | 0 | 1 | 1 | 20
  Not on Metformin, But On At Least 2 Other Medications | 0 | 0 | 3 | 2 | 0 | 2 | 1 | 1 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of HbA1C (Glycated Hemoglobin)
Description: Least Squares Means change in HbA1C from baseline to Week 12 of the treatment period, where HbA1C is reported in units of percent. The change in HbA1c from baseline to Week 12 is expressed as a change in the value of HbA1C.
Time Frame: baseline (Run-in period, Week 0, Visit 1) and Week 12 (follow-up)
Population: Data collected from participants who received excipient-matched placebo was an exploratory efficacy evaluation and therefore excluded from the primary and secondary analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent HbA1C
Groups:
- Combined Cohort A +Cohort B: Matched-Placebo Oral Capsule: Placebo matched to one of the three active comparator arms. (either QHS, BID, or TID)
  Placebo oral capsule: Placebo provided QHS, BID, TID
  Data collected from participants who received excipient-matched placebo was an exploratory efficacy evaluation and therefore excluded from the primary and secondary analysis.
Arm/Group | Combined Cohort A +Cohort B: Matched-Placebo Oral Capsule | Cohort A: ORMD-0801 Once Daily - QHS | Cohort A: ORMD-0801 Twice Daily - BID | Cohort A: ORMD-0801 Three Times Daily - TID | Cohort B:ORMD-0801, 8 mg Once Daily - QHS: | Cohort B: ORMD-0801 8 mg Twice Daily - BID | Cohort B: ORMD-0801 16 mg Once Daily - QHS: | Cohort B: ORMD-0801 16 mg Twice Daily - BID
Number analyzed (Participants) | 53 | 59 | 54 | 52 | 13 | 12 | 13 | 10
percent HbA1C | -0.13 [-0.86 to 0.59] | -0.60 [-1.37 to 0.16] | -0.59 [-1.32 to 0.14] | -0.51 [-1.27 to 0.25] | -0.95 [-1.87 to -0.03] | -0.95 [-1.84 to -0.07] | 0.12 [-0.80 to 1.04] | -0.50 [-1.47 to 0.48]

2. Secondary Outcome: Mean Change From Baseline Over Time for HbA1C
Description: Mean change from baseline (Run-In, Week 0 Visit 1) to Part 1, Visit 3 for HbA1C (measured in mmols/mol)
Time Frame: Baseline (Run-In:Week 0, Visit 1) to Part 1, Visit 3, elapsed time: 3 weeks.
Population: Intend-to-Treat; data collected from participants who received excipient-matched placebo was an exploratory efficacy evaluation and therefore excluded from the primary and secondary analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/mol
Groups:
- Combined Cohort A+Cohort B: Matched-Placebo Oral Capsule: Placebo matched to one of the three active comparator arms. (either QHS, BID, or TID)
  Placebo oral capsule: Placebo provided QHS, BID, TID
  Data collected from participants who received excipient-matched placebo was an exploratory efficacy evaluation and therefore excluded from the primary and secondary analysis.
Arm/Group | Combined Cohort A+Cohort B: Matched-Placebo Oral Capsule | Cohort A: ORMD-0801 Once Daily - QHS | Cohort A: ORMD-0801 Twice Daily - BID | Cohort A: ORMD-0801 Three Times Daily - TID | Cohort B:ORMD-0801, 8 mg Once Daily - QHS: | Cohort B: ORMD-0801 8 mg Twice Daily - BID | Cohort B: ORMD-0801 16 mg Once Daily - QHS: | Cohort B: ORMD-0801 16 mg Twice Daily - BID
Number analyzed (Participants) | 61 | 62 | 62 | 58 | 14 | 13 | 14 | 14
mmol/mol | -2.12 [-4.40 to 0.16] | -2.56 [-4.94 to -0.19] | -1.95 [-4.21 to 0.30] | -2.91 [-5.25 to -0.57] | -3.26 [-6.13 to -0.39] | -5.51 [-8.30 to -2.73] | -2.06 [-4.94 to 0.82] | -1.87 [-4.72 to 0.98]

3. Secondary Outcome: Change Over Time in Hb1Ac
Description: Change of Hb1Ac from Baseline to Week 10, measured in mmol/mol
Time Frame: Baseline (week 0, visit 1) to Week 10, part 2
Population: Intent-to-Treat; data collected from participants who received excipient-matched placebo was an exploratory efficacy evaluation and therefore excluded from the primary and secondary analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/mol
Groups:
- Cohort A+Cohort B: Combined Matched Placebo Oral Capsule: Placebo matched to one of the three active comparator arms. (either QHS, BID, or TID)
  Placebo oral capsule: Placebo provided QHS, BID, TID
  Data collected from participants who received excipient-matched placebo was an exploratory efficacy evaluation and therefore excluded from the primary and secondary analysis.
Arm/Group | Cohort A+Cohort B: Combined Matched Placebo Oral Capsule | Cohort A: ORMD-0801 Once Daily - QD | Cohort A: ORMD-0801 Twice Daily - BID | Cohort A: ORMD-0801 Three Times Daily - TID | Cohort B:ORMD-0801, 8 mg Once Daily - QD | Cohort B: ORMD-0801 8 mg Twice Daily - BID | Cohort B: ORMD-0801 16 mg Once Daily - QD | Cohort B: ORMD-0801 16 mg Twice Daily - BID
Number analyzed (Participants) | 53 | 58 | 54 | 50 | 13 | 12 | 13 | 11
mmol/mol | -1.27 [-8.88 to 6.35] | -5.95 [-14.05 to 2.16] | -4.95 [-12.62 to 2.73] | -6.16 [-14.22 to 1.90] | -10.34 [-20.01 to -0.68] | -10.71 [-20.02 to -1.40] | -0.25 [-9.94 to 9.44] | -4.66 [-14.61 to 5.28]

ADVERSE EVENTS:
Time Frame: Each subject was followed for a period of 12 weeks
Description: Data collected from participants who received excipient matched placebo was an exploratory efficacy evaluation and therefore excluded from the primary and secondary analysis.
Groups:
- Combined Cohort A + Cohort B: Matched Placebo: Placebo matched to one of the three active comparator arms. (either QHS, BID, or TID)
  Placebo oral capsule: Placebo provided QHS, BID, TID
  Per FDA, the sub-Cohort A, excipient-matched placebo TID is an exploratory arm and is not part of the primary analysis.
- Excipient Matched Placebo -TID: Exploratory endpoint not part of primary analysis per FDA
Arm/Group | Combined Cohort A + Cohort B: Matched Placebo | Cohort A: ORMD-0801 Once Daily - QD | Cohort A: ORMD-0801 Twice Daily - BID | Cohort A: ORMD-0801 Three Times Daily - TID | Cohort B:ORMD-0801, 8 mg Once Daily - QD | Cohort B: ORMD-0801 8 mg Twice Daily - BID | Cohort B: ORMD-0801 16 mg Once Daily - QD | Cohort B: ORMD-0801 16 mg Twice Daily - BID | Excipient Matched Placebo -TID
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/69 | 0/68 | 0/69 | 0/15 | 0/17 | 0/18 | 0/15 | 1/20
Serious Adverse Events (participants affected / at risk) | 0/82 | 5/69 | 0/68 | 3/69 | 0/15 | 0/17 | 0/18 | 1/15 | 3/20
Other Adverse Events (participants affected / at risk) | 11/82 | 19/69 | 6/68 | 10/69 | 5/15 | 2/17 | 1/18 | 2/15 | 13/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Cohort A + Cohort B: Matched Placebo (N=82) | Cohort A: ORMD-0801 Once Daily - QD (N=69) | Cohort A: ORMD-0801 Twice Daily - BID (N=68) | Cohort A: ORMD-0801 Three Times Daily - TID (N=69) | Cohort B:ORMD-0801, 8 mg Once Daily - QD (N=15) | Cohort B: ORMD-0801 8 mg Twice Daily - BID (N=17) | Cohort B: ORMD-0801 16 mg Once Daily - QD (N=18) | Cohort B: ORMD-0801 16 mg Twice Daily - BID (N=15) | Excipient Matched Placebo -TID (N=20)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Cohort A + Cohort B: Matched Placebo (N=82) | Cohort A: ORMD-0801 Once Daily - QD (N=69) | Cohort A: ORMD-0801 Twice Daily - BID (N=68) | Cohort A: ORMD-0801 Three Times Daily - TID (N=69) | Cohort B:ORMD-0801, 8 mg Once Daily - QD (N=15) | Cohort B: ORMD-0801 8 mg Twice Daily - BID (N=17) | Cohort B: ORMD-0801 16 mg Once Daily - QD (N=18) | Cohort B: ORMD-0801 16 mg Twice Daily - BID (N=15) | Excipient Matched Placebo -TID (N=20)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Atrioventricular Block First Degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 3 (3) | 8 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Large Intestine Polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic Cyst (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal Allergy (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenoviral upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body Tinea (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dispepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atypical Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mulscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal Discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracardiac Mass (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/32/NCT03467932/Prot_SAP_000.pdf